CLINICAL TRIAL: NCT02653703
Title: High-concentration L-menthol as a Counter-irritant to TRPA1-induced Neurogenic Inflammation, Thermal and Mechanical Hyperalgesia Caused by Trans-cinnamaldehyde
Brief Title: L-menthol as a Topical Counter-irritant to TRPA1-induced Neurogenic Inflammation and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Parisa Gazerani, Professor, PharmD, Ph.D., Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: N-20130005
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Inflammation; Pruritus; Hyperalgesia
MeSH Terms: conditions — Inflammation; Pruritus; Hyperalgesia | interventions — Menthol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle, topical ethanol 96% (Placebo Comparator): Exposure: 10 % topical trans-cinnamaldehyde [CAS Number: 14371-10-9] Vehicle: 96% ethanol
  Interventions: Other: Vehicle, topical ethanol 96%
- Topical L-menthol 40% (Experimental): Exposure: 10 % trans-cinnamaldehyde [CAS Number: 14371-10-9] Intervention: 40% l-menthol [CAS Number: 2216-51-5] Vehicle: 96% ethanol
  Interventions: Other: Topical L-menthol 40%

INTERVENTIONS:
Other: Topical L-menthol 40% — Naturally occurring local anaesthetic, counterirritant and TPRM8-agonist. CAS Number: 2216-51-5
  Other Names: Menthol
  Arms: Topical L-menthol 40%
Other: Vehicle, topical ethanol 96% — Organic solvent CAS Number: 64-17-5
  Arms: Vehicle, topical ethanol 96%

SUMMARY:
The aim of this study is to quantitatively characterize the effects of L-menthol as a topical counter-irritant on cutaneous pain and hyperalgesia provoked by topical application of the TRPA1-agonist trans-cinnamaldehyde (CA) in healthy human volunteers.

DETAILED DESCRIPTION:
This study is designed as an experimental model in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* 18 healthy men and women aged 18-50 years willing to abstain from alcohol, nicotine, caffeine and pain medication 24 hours before experimental sessions

Exclusion Criteria:

* Pregnancy
* Skin disorders (e.g. contact eczema)
* Chronic pain conditions
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate

Ages: 18 Years to 50 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Spontaneous pain intensity [self-reported on a visual analog scale] | 0-20 minutes with a sampling frequency of 1/1 min
  Rating of the overall pain intensity on a visual analog scale (VAS ranging from "No pain" = 0, to "worst imaginable pain" =10) once every minute

SECONDARY OUTCOMES:
Neurogenic inflammation [Measured by Laser speckle flowmetry in a 3x3 cm area] | 20-25 minutes post induction
  Speckle contrast flowmetry (MoorFLPI, Moor Instruments, Devon, UK). The assessment is conducted with a 30-cm distance between the head of the laser and the application area with an exposure time of 8.3ms. Single frame images are analyzed on appertaining software (MoorFLPI Review V 4.0, Moor Instruments), upon which the arithmetic mean flux (arbitrary units) is calculated. The longitudinal analysis of the spatial dispersion of neurogenic inflammation is performed using the line histogram tool. A 7-cm line centered in the area of application was placed longitudinally along the volar forearm and the perfusion intensity is recorded every 2.5 mm.
Heat hyperalgesia | 25-27.5 minutes post induction
  Heat pain threshold assessments is performed with a Medoc Pathway (Medoc Ltd, Ramat Yishay, Israel) equipped with a 3 × 3 cm advanced thermal stimulator probe where the baseline temperature was set to 32 °C. Ramp stimuli of 1 °C/s are delivered and the subjects are asked to identify the heat pain threshold upon which the temperature is returned to the baseline at a rate of 5 °C/s. The test result is calculated as the arithmetic mean of the outcome from three repeated stimuli. Heat hyperalgesia is considered to be a significant drop in heat pain threshold
Mechanical hyperalgesia | 27.5-30 minutes post induction
  To evaluate the mechanical pain threshold (MPT) an electronic von Frey transducer and an electronic coVAS connected to a SENSE-Box setup is used (both items: Somedic, Hörby, Sweden). Five ramp stimuli from 0-110 g at a rate of 5g/1 sec with the default stimulus probe is conducted at different locations within the application area. The subjects are instructed to continuously rate the perceived pain on the coVAS ranging from "No pain" (0) to "worst imaginable pain" (10). The arithmetic mean of the VAS scores yields three MPTs (fixed to VAS = 0.5, 1 and 2) and an area-under-the-curve (AUC).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Olsen RV, Andersen HH, Moller HG, Eskelund PW, Arendt-Nielsen L. Somatosensory and vasomotor manifestations of individual and combined stimulation of TRPM8 and TRPA1 using topical L-menthol and trans-cinnamaldehyde in healthy volunteers. Eur J Pain. 2014 Oct;18(9):1333-42. doi: 10.1002/j.1532-2149.2014.494.x. Epub 2014 Mar 25. PMID 24664788
- [Background] Hojland CR, Andersen HH, Poulsen JN, Arendt-Nielsen L, Gazerani P. A human surrogate model of itch utilizing the TRPA1 agonist trans-cinnamaldehyde. Acta Derm Venereol. 2015 Sep;95(7):798-803. doi: 10.2340/00015555-2103. PMID 25792226
- [Background] Namer B, Seifert F, Handwerker HO, Maihofner C. TRPA1 and TRPM8 activation in humans: effects of cinnamaldehyde and menthol. Neuroreport. 2005 Jun 21;16(9):955-9. doi: 10.1097/00001756-200506210-00015. PMID 15931068
- [Background] Namer B, Kleggetveit IP, Handwerker H, Schmelz M, Jorum E. Role of TRPM8 and TRPA1 for cold allodynia in patients with cold injury. Pain. 2008 Sep 30;139(1):63-72. doi: 10.1016/j.pain.2008.03.007. Epub 2008 Apr 25. PMID 18440147
- [Background] Andersen HH, Olsen RV, Moller HG, Eskelund PW, Gazerani P, Arendt-Nielsen L. A review of topical high-concentration L-menthol as a translational model of cold allodynia and hyperalgesia. Eur J Pain. 2014 Mar;18(3):315-25. doi: 10.1002/j.1532-2149.2013.00380.x. Epub 2013 Aug 20. PMID 23963768
- [Background] Leslie TA, Greaves MW, Yosipovitch G. Current topical and systemic therapies for itch. Handb Exp Pharmacol. 2015;226:337-56. doi: 10.1007/978-3-662-44605-8_18. PMID 25861788
- [Background] Heyneman CA. Topical nonsteroidal antiinflammatory drugs for acute soft tissue injuries. Ann Pharmacother. 1995 Jul-Aug;29(7-8):780-2. doi: 10.1177/106002809502907-822. PMID 8520097
- [Derived] Andersen HH, Gazerani P, Arendt-Nielsen L. High-Concentration L-Menthol Exhibits Counter-Irritancy to Neurogenic Inflammation, Thermal and Mechanical Hyperalgesia Caused by Trans-cinnamaldehyde. J Pain. 2016 Aug;17(8):919-29. doi: 10.1016/j.jpain.2016.05.004. Epub 2016 May 31. PMID 27260636